CLINICAL TRIAL: NCT03718585
Title: Whole Exome Sequencing Analysis Project in Chronic Kidney Disease Patients With Nocturnal Hypertension
Brief Title: Whole Exome Sequencing in CKD Hypertension
Acronym: WESCH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Cheng Wang, Director of Nephrology, Fifth Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: ZDWY.SNK.001
Record Dates: First submitted 2018-10-23; First posted 2018-10-24 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Hypertension;Nephropathy
Keywords: Nocturnal Hypertension; Chronic Kidney Disease; Whole Exome Sequencing
MeSH Terms: conditions — Hypertensive Nephropathy; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- nocturnal group: Chronic kidney disease patients with nocturnal hypertension
  Interventions: Other: whole exome sequencing analysis
- non-nocturnal group: Chronic kidney disease patients without nocturnal hypertension
  Interventions: Other: whole exome sequencing analysis
- non-CKD group: patients without chronic kidney disease
  Interventions: Other: whole exome sequencing analysis

INTERVENTIONS:
Other: whole exome sequencing analysis — Collecting peripheral blood samples (2 ml) from subjects for whole exome sequencing

SUMMARY:
The prevalence of hypertension in patients with CKD in China is high but the control rate is low. Compared with the single blood pressure measurement method of the blood pressure of the office, ambulatory blood pressure monitoring (ABPM) can reflect the overall situation of 24-hour blood pressure, dynamic fluctuation degree and circadian rhythm change more completely and objectively. Studies have shown that patients with CKD with hypertension have their own uniqueness through ABPM measurement, and nocturnal hypertension is the main cause of poor blood pressure control. Further studies have shown that nocturnal hypertension is an independent and more effective prognostic indicator of death and CVD in patients with hypertension. Evidence from European and American countries suggests that in the CKD population, elevated nighttime blood pressure is more predictive of CKD progression or CVD than daytime blood pressure. Compared with countries such as Europe and the United States, there are differences in the causes, genetic background and daily behaviors of kidney disease in our population. It is urgent to investigate the predictive value of nocturnal hypertension for renal end point and CVD in CKD population in China. To this end, our study found for the first time that CKD patients generally have changes in nocturnal blood pressure patterns, and the anti-dope type blood pressure pattern is closely related to the target organ damage. Our further study found that the incidence of nocturnal hypertension in Chinese patients with CKD is more than 50%, and compared with non-dipping blood pressure, patients with nocturnal hypertension have more serious target organ damage, which is independent risk factors for all-cause death, cardiovascular death, renal events, and cardiovascular events in patients with CKD. These preliminary results suggest the role of nocturnal hypertension in the prognosis of CKD patients in China, but there are still the following questions: Is the occurrence of nocturnal hypertension in CKD patients related to certain gene expression? This project intends to perform whole-genome exon sequencing and analysis on CKD patients with nocturnal hypertension to determine the genetic mechanism of CKD patients with nocturnal hypertension. The completion of the subject will reveal the genetic characteristics of CKD patients with nocturnal hypertension, and provide a basis for the precise prevention and treatment of chronic kidney disease hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 14 years old and <75years.
2. The clinical data during the hospitalization period are detailed and complete.
3. Follow-up information is available.
4. Ambulatory blood pressure monitoring indicates nighttime blood pressure SBP≥120mmHg and/or DBP≥70mmHg.
5. Diagnosed as CKD according to the 2012 KDIGO guidelines, abnormalities of kidney structure or function, present for >3 months, with implications for health, including glomerular filtration rate (GFR) normal and abnormal pathological damage, blood (abnormal electrolyte or other components caused by renal tubular dysfunction) or urine components (proteinuria: ACR ≥ 30mg / gCr; other abnormal urine components) abnormal, and imaging abnormalities; or unexplained GFR decline (< 60 ml/min/1.73 m2); and eGFR ≥ 30 ml/min/1.73 m2.

Exclusion Criteria:

1. pregnancy.
2. combined tumors.
3. There is a history of drug abuse or alcohol abuse.
4. There are serious infections recently.
5. Life expectancy is less than half a year.
6. Renal replacement therapy has been performed.
7. Acquired immunodeficiency syndrome.
8. Those who are being treated with cortisol hormones.
9. Those who study or work at night for a long time and have irregular rest.
10. Those who cannot cooperate or are unable to tolerate ambulatory blood pressure monitors.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
whole exome sequencing analysis | 4 years
  Collecting peripheral blood samples (2 ml) from subjects for whole exome sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Wang, Director, Principal Investigator — Nephrology Department, the Fifth Affiliated Hospital of Sun Yat-sen University
Locations (1):
- Fifth Affiliated Hospital, Sun Yat-Sen University, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ricardo AC, Flessner MF, Eckfeldt JH, Eggers PW, Franceschini N, Go AS, Gotman NM, Kramer HJ, Kusek JW, Loehr LR, Melamed ML, Peralta CA, Raij L, Rosas SE, Talavera GA, Lash JP. Prevalence and Correlates of CKD in Hispanics/Latinos in the United States. Clin J Am Soc Nephrol. 2015 Oct 7;10(10):1757-66. doi: 10.2215/CJN.02020215. Epub 2015 Sep 28. PMID 26416946
- [Background] Zhang L, Wang F, Wang L, Wang W, Liu B, Liu J, Chen M, He Q, Liao Y, Yu X, Chen N, Zhang JE, Hu Z, Liu F, Hong D, Ma L, Liu H, Zhou X, Chen J, Pan L, Chen W, Wang W, Li X, Wang H. Prevalence of chronic kidney disease in China: a cross-sectional survey. Lancet. 2012 Mar 3;379(9818):815-22. doi: 10.1016/S0140-6736(12)60033-6. PMID 22386035
- [Background] Foley RN. Clinical epidemiology of cardiovascular disease in chronic kidney disease. J Ren Care. 2010 May;36 Suppl 1:4-8. doi: 10.1111/j.1755-6686.2010.00171.x. PMID 20586894
- [Background] Wang C, Ye Z, Li Y, Zhang J, Zhang Q, Ma X, Peng H, Lou T. Prognostic Value of Reverse Dipper Blood Pressure Pattern in Chronic Kidney Disease Patients not Undergoing Dialysis: Prospective Cohort Study. Sci Rep. 2016 Oct 7;6:34932. doi: 10.1038/srep34932. PMID 27713498
- [Background] Pogue V, Rahman M, Lipkowitz M, Toto R, Miller E, Faulkner M, Rostand S, Hiremath L, Sika M, Kendrick C, Hu B, Greene T, Appel L, Phillips RA; African American Study of Kidney Disease and Hypertension Collaborative Research Group. Disparate estimates of hypertension control from ambulatory and clinic blood pressure measurements in hypertensive kidney disease. Hypertension. 2009 Jan;53(1):20-7. doi: 10.1161/HYPERTENSIONAHA.108.115154. Epub 2008 Dec 1. PMID 19047584
- [Background] Global Burden of Metabolic Risk Factors for Chronic Diseases Collaboration. Cardiovascular disease, chronic kidney disease, and diabetes mortality burden of cardiometabolic risk factors from 1980 to 2010: a comparative risk assessment. Lancet Diabetes Endocrinol. 2014 Aug;2(8):634-47. doi: 10.1016/S2213-8587(14)70102-0. Epub 2014 May 16. PMID 24842598
- [Background] Wang C, Deng WJ, Gong WY, Zhang J, Zhang QZ, Ye ZC, Lou T. Nocturnal Hypertension Correlates Better With Target Organ Damage in Patients With Chronic Kidney Disease than a Nondipping Pattern. J Clin Hypertens (Greenwich). 2015 Oct;17(10):792-801. doi: 10.1111/jch.12589. Epub 2015 Jun 4. PMID 26041362
- [Background] Zheng Y, Cai GY, Chen XM, Fu P, Chen JH, Ding XQ, Yu XQ, Lin HL, Liu J, Xie RJ, Wang LN, Ni ZH, Liu FY, Yin AP, Xing CY, Wang L, Shi W, Liu JS, He YN, Ding GH, Li WG, Wu GL, Miao LN, Chen N, Su Z, Mei CL, Zhao JY, Gu Y, Bai YK, Luo HM, Lin S, Chen MH, Gong L, Yang YB, Yang XP, Li Y, Wan JX, Wang NS, Li HY, Xi CS, Hao L, Xu Y, Fang JA, Liu BC, Li RS, Wang R, Zhang JH, Wang JQ, Lou TQ, Shao FM, Mei F, Liu ZH, Yuan WJ, Sun SR, Zhang L, Zhou CH, Chen QK, Jia SL, Gong ZF, Guan GJ, Xia T, Zhong LB; Prevalence, Awareness, and Treatment Rates in Chronic Kidney Disease Patients with Hypertension in China (PATRIOTIC) Collaborative Group. Prevalence, awareness, treatment, and control of hypertension in the non-dialysis chronic kidney disease patients. Chin Med J (Engl). 2013 Jun;126(12):2276-80. PMID 23786938
- [Background] Luan FL, Norman SP. Intensive blood-pressure control in hypertensive chronic kidney disease. N Engl J Med. 2010 Dec 23;363(26):2564-5; author reply 2565-6. doi: 10.1056/NEJMc1011419. No abstract available. PMID 21175325
- [Background] O'Brien E, Sheridan J, O'Malley K. Dippers and non-dippers. Lancet. 1988 Aug 13;2(8607):397. doi: 10.1016/s0140-6736(88)92867-x. No abstract available. PMID 2899801
- [Background] Hodgkinson J, Mant J, Martin U, Guo B, Hobbs FD, Deeks JJ, Heneghan C, Roberts N, McManus RJ. Relative effectiveness of clinic and home blood pressure monitoring compared with ambulatory blood pressure monitoring in diagnosis of hypertension: systematic review. BMJ. 2011 Jun 24;342:d3621. doi: 10.1136/bmj.d3621. PMID 21705406
- [Background] Mancia G, Fagard R, Narkiewicz K, Redon J, Zanchetti A, Bohm M, Christiaens T, Cifkova R, De Backer G, Dominiczak A, Galderisi M, Grobbee DE, Jaarsma T, Kirchhof P, Kjeldsen SE, Laurent S, Manolis AJ, Nilsson PM, Ruilope LM, Schmieder RE, Sirnes PA, Sleight P, Viigimaa M, Waeber B, Zannad F; Task Force for the Management of Arterial Hypertension of the European Society of Hypertension and the European Society of Cardiology. 2013 ESH/ESC Practice Guidelines for the Management of Arterial Hypertension. Blood Press. 2014 Feb;23(1):3-16. doi: 10.3109/08037051.2014.868629. Epub 2013 Dec 20. No abstract available. PMID 24359485
- [Background] ESH/ESC Task Force for the Management of Arterial Hypertension. 2013 Practice guidelines for the management of arterial hypertension of the European Society of Hypertension (ESH) and the European Society of Cardiology (ESC): ESH/ESC Task Force for the Management of Arterial Hypertension. J Hypertens. 2013 Oct;31(10):1925-38. doi: 10.1097/HJH.0b013e328364ca4c. No abstract available. PMID 24107724
- [Background] Mojon A, Ayala DE, Pineiro L, Otero A, Crespo JJ, Moya A, Boveda J, de Lis JP, Fernandez JR, Hermida RC; Hygia Project Investigators. Comparison of ambulatory blood pressure parameters of hypertensive patients with and without chronic kidney disease. Chronobiol Int. 2013 Mar;30(1-2):145-58. doi: 10.3109/07420528.2012.703083. Epub 2012 Oct 25. PMID 23181690
- [Background] Yano Y, Kario K. Nocturnal blood pressure and cardiovascular disease: a review of recent advances. Hypertens Res. 2012 Jul;35(7):695-701. doi: 10.1038/hr.2012.26. Epub 2012 Mar 1. PMID 22378470
- [Background] Clement DL, De Buyzere ML, De Bacquer DA, de Leeuw PW, Duprez DA, Fagard RH, Gheeraert PJ, Missault LH, Braun JJ, Six RO, Van Der Niepen P, O'Brien E; Office versus Ambulatory Pressure Study Investigators. Prognostic value of ambulatory blood-pressure recordings in patients with treated hypertension. N Engl J Med. 2003 Jun 12;348(24):2407-15. doi: 10.1056/NEJMoa022273. PMID 12802026
- [Background] Hermida RC. Sleep-time ambulatory blood pressure as a prognostic marker of vascular and other risks and therapeutic target for prevention by hypertension chronotherapy: Rationale and design of the Hygia Project. Chronobiol Int. 2016;33(7):906-36. doi: 10.1080/07420528.2016.1181078. Epub 2016 May 24. PMID 27221952
- [Background] Hermida RC, Ayala DE, Smolensky MH, Fernandez JR, Mojon A, Portaluppi F. Chronotherapy with conventional blood pressure medications improves management of hypertension and reduces cardiovascular and stroke risks. Hypertens Res. 2016 May;39(5):277-92. doi: 10.1038/hr.2015.142. Epub 2015 Dec 10. PMID 26657008
- [Background] Hermida RC, Ayala DE, Mojon A, Fernandez JR. Bedtime dosing of antihypertensive medications reduces cardiovascular risk in CKD. J Am Soc Nephrol. 2011 Dec;22(12):2313-21. doi: 10.1681/ASN.2011040361. Epub 2011 Oct 24. PMID 22025630
- [Background] Hermida RC, Ayala DE, Mojon A, Fernandez JR. Decreasing sleep-time blood pressure determined by ambulatory monitoring reduces cardiovascular risk. J Am Coll Cardiol. 2011 Sep 6;58(11):1165-73. doi: 10.1016/j.jacc.2011.04.043. PMID 21884956
- [Background] Hansen TW, Li Y, Boggia J, Thijs L, Richart T, Staessen JA. Predictive role of the nighttime blood pressure. Hypertension. 2011 Jan;57(1):3-10. doi: 10.1161/HYPERTENSIONAHA.109.133900. Epub 2010 Nov 15. PMID 21079049
- [Background] Felicio JS, de Souza AC, Kohlmann N, Kohlmann O Jr, Ribeiro AB, Zanella MT. Nocturnal blood pressure fall as predictor of diabetic nephropathy in hypertensive patients with type 2 diabetes. Cardiovasc Diabetol. 2010 Aug 13;9:36. doi: 10.1186/1475-2840-9-36. PMID 20704750
- [Background] Redon J, Plancha E, Swift PA, Pons S, Munoz J, Martinez F. Nocturnal blood pressure and progression to end-stage renal disease or death in nondiabetic chronic kidney disease stages 3 and 4. J Hypertens. 2010 Mar;28(3):602-7. doi: 10.1097/HJH.0b013e328333fe4d. PMID 20150824
- [Background] Mehta R, Drawz PE. Is nocturnal blood pressure reduction the secret to reducing the rate of progression of hypertensive chronic kidney disease? Curr Hypertens Rep. 2011 Oct;13(5):378-85. doi: 10.1007/s11906-011-0217-8. PMID 21710375
- [Background] Wang C, Zhang J, Liu X, Li C, Ye Z, Peng H, Chen Z, Lou T. Reversed dipper blood-pressure pattern is closely related to severe renal and cardiovascular damage in patients with chronic kidney disease. PLoS One. 2013;8(2):e55419. doi: 10.1371/journal.pone.0055419. Epub 2013 Feb 5. PMID 23393577